CLINICAL TRIAL: NCT05482256
Title: The Role of Detergents in the Pathogenesis of Eosinophilic Esophagitis
Brief Title: A Study of Detergents in the Pathogenesis of Eosinophilic Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin L. Wright, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-003963
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Sodium Fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toothpaste detergents with Eosinophilic Esophagitis Testing (Experimental): Subjects will complete an esophageal string test prior to and after completing a high resolution esophageal manometry then brushing their teeth using Colgate toothpaste.
  Interventions: Diagnostic Test: Esophageal String Test (EST); Other: Colgate; Diagnostic Test: High Resolution Esophageal Manometry (HREM)

INTERVENTIONS:
Diagnostic Test: Esophageal String Test (EST) — Non-invasive, FDA-registered sampling method to evaluate eosinophilic inflammation in the esophagus. The EST is performed by having an individual swallow a capsule attached to a string which captures secretions from the esophagus. The end of the string is taped to the cheek and the capsule is swallowed with water. After 1 hour, the EST will be removed, and the string will be processed for laboratory analysis.
  Other Names: EnteroTracker
Other: Colgate — 2 grams of toothpaste (pea sized amount) for 2 minutes
Diagnostic Test: High Resolution Esophageal Manometry (HREM) — Thin flexible tube with sensors placed in the nose and swallowed for esophagus placement to conduct reading regarding the lining of the esophagus taken for approximately 10 minutes

SUMMARY:
The purpose of this research is to determine if detergents in everyday products such as toothpaste make the lining of the esophagus leaky and cause allergic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy volunteers.
* Able to swallow pills.

Exclusion Criteria:

* Personal history of esophageal disease including but not limited to eosinophilic esophagitis, esophageal dysmotility, or GERD/reflux.
* History of dysphagia (i.e., difficulty swallowing), chronic vomiting, chronic abdominal pain, unintentional weight loss.
* Celiac disease, inflammatory bowel disease, irritable bowel syndrome, esophageal varices, chronic aspiration, connective tissue disorder, or known parasitic infection.
* Gelatin allergy.
* Use of a toothpaste containing SLS within 2 weeks of the study.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Change in Mucosal impedance 15 minutes after exposure | Baseline, 15 minutes after teeth brushing
  Recorded from the High Resolution Esophageal Manometry testing that measures eosinophils on histology

SECONDARY OUTCOMES:
Change in Mucosal impedance 30 minutes after exposure | Baseline, 30 minutes after teeth brushing
  Recorded from the High Resolution Esophageal Manometry testing that measures eosinophils on histology
Change in Mucosal impedance 45 minutes after exposure | Baseline, 45 minutes after teeth brushing
  Recorded from the High Resolution Esophageal Manometry testing that measures eosinophils on histology
Change in Mucosal impedance 60 minutes after exposure | Baseline, 60 minutes after teeth brushing
  Recorded from the High Resolution Esophageal Manometry testing that measures eosinophils on histology
Change in IL-33 levels | Baseline, approximately 60 minutes after teeth brushing
  Measured from esophageal string test eluates

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Wright, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic - Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20535089